CLINICAL TRIAL: NCT01260363
Title: Pain Treatment After Anterior Cruciate Ligament Reconstruction
Brief Title: Comparison of Infiltration Analgesia With Femoral Nerve Block After Hamstrings Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-022500-50
Record Dates: First submitted 2010-12-06; First posted 2010-12-15 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Injury of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naropin, Adrenalin, applicationsite (Active Comparator)
  Interventions: Procedure: Local infiltration analgesia
- Femoral nerve block (Active Comparator)
  Interventions: Procedure: Femoral nerve block

INTERVENTIONS:
Procedure: Femoral nerve block — Femoral nerve block ultrasound guidet with ropivacaine 20ml 2.5mg/ml
  Other Names: FNB
  Arms: Femoral nerve block
Procedure: Local infiltration analgesia — Local infiltration analgesia with ropivacaine 2.5mg/ml with epfinedrine 5mikrogram/ml. 20ml at harvest site and 20ml at incisionsites.
  Other Names: LIA teknik
  Arms: Naropin, Adrenalin, applicationsite

SUMMARY:
Pain treatment after anterior cruciate ligament reconstruction - Comparison of infiltration analgesia with femoral nerve block after.

DETAILED DESCRIPTION:
Inclusion Criteria:

* Patients undergoing primary anetrior cruciate ligament reconstruction with semiTendinos/gracillis graft
* Age > 18 year

Exclusion Criteria:

* Revision ACL reconstruction
* Patients with cartilige lision
* Patients with arthritis
* Pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary anetrior cruciate ligament reconstruction with semiTendinos/gracillis graft
* Age > 18 year

Exclusion Criteria:

* Revision ACL reconstruction
* Patients with cartilige lision
* Patients with arthritis
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Numeric Rang Scale pain | 1 day after operation

SECONDARY OUTCOMES:
use of analgetics | 0h, 3h, 24h, 48h

CONTACTS AND LOCATIONS:
Overall Officials: Theis Thillemann, MD, Ph.d., Principal Investigator — Regional hospital Horsens, Denmark
Locations (1):
- Regional Hospital Horsens, Horsens, Denmark

REFERENCES:
- [Derived] Kristensen PK, Pfeiffer-Jensen M, Storm JO, Thillemann TM. Local infiltration analgesia is comparable to femoral nerve block after anterior cruciate ligament reconstruction with hamstring tendon graft: a randomised controlled trial. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):317-23. doi: 10.1007/s00167-013-2399-x. Epub 2013 Jan 23. PMID 23338666